CLINICAL TRIAL: NCT04016324
Title: InterStim Basic Evaluation Lead Post Market Clinical Follow-Up Study
Brief Title: InterStim Basic Evaluation Lead Post-Market Clinical Follow-up Study
Acronym: BASIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT19002
Record Dates: First submitted 2019-07-09; First posted 2019-07-11 (Actual); Results first posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Overactive Bladder; Urinary Urge Incontinence; Urgency-frequency Syndrome
Keywords: Overactive Bladder; Urinary Urge Incontinence; Urgency-frequency Syndrome
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge

STUDY DESIGN:
Intervention Model Description: To characterize proportion of subjects who demonstrate motor or sensory response(s) during lead placement using the InterStim Basic Evaluation Lead.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Basic evaluation (Other): Subjects with overactive bladder will go through InterStim basic evaluation with the commercially approved foramen needle and basic evaluation kit.
  Interventions: Device: InterStim Basic Evaluation lead and foramen needle

INTERVENTIONS:
Device: InterStim Basic Evaluation lead and foramen needle — Commercial devices within their intended use as described in approved Instructions for Use.

SUMMARY:
Post-market clinical follow-up for continued assessment of safety and performance of the InterStim basic evaluation lead and foramen needle(s) used during a therapy evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 years of age or older
2. Candidate for sacral neuromodulation in accordance with the InterStim System labeling
3. Have a diagnosis of overactive bladder (OAB) as demonstrated by either urinary urge incontinence and/or urinary frequency on a 3-day voiding diary
4. Willing and able to accurately complete study diaries, questionnaire, attend visits, and comply with the study protocol
5. Willing and able to provide signed and dated informed consent

Exclusion Criteria:

1. Have neurological conditions such as multiple sclerosis, clinically significant peripheral neuropathy or spinal cord injury (e.g., paraplegia)
2. Have implantable pacemakers, or defibrillators
3. Have primary stress incontinence or mixed incontinence where the stress component overrides the urge component
4. Have knowledge of planned MRIs, diathermy, microwave exposure, high output ultrasonic exposure, or radio frequency (RF) energy exposure not included within the scanning conditions provided with the InterStim System labeling
5. Women who are pregnant or planning to become pregnant during participation in the study
6. Characteristics indicating a poor understanding of the study or characteristics that indicate the subject may have poor compliance with the study protocol requirements
7. Concurrent participation in another clinical study that may add additional safety risks and/or confound study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: BASIC Clinical Research Study Team, Study Director — Medtronic
Locations (15):
- United States (10):
  - Pinellas Urology, St. Petersburg, Florida
  - Florida Urology Partners, Tampa, Florida
  - Minnesota Urology (Plymouth), Plymouth, Minnesota
  - Urologic Research and Consulting, Englewood, New Jersey
  - FirstHealth Urogynecology, Hamlet, North Carolina
  - Wright State Physicians, Fairborn, Ohio
  - Prisma Health, Greenville, South Carolina
  - Southern Urogynecology, West Columbia, South Carolina
  - Urology Partners of North Texas, Arlington, Texas
  - Urology of Virginia, Virginia Beach, Virginia
- University Urology Associates, Toronto, Ontario, Canada
- Radboud UMC, Nijmegen, Netherlands
- United Kingdom (3):
  - The Bristol Urological Institute, Bristol
  - The Newcastle upon Tyne Hospitals, Newcastle upon Tyne
  - Salford Royal NHS Foundation Trust, Salford

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were considered to be 'enrolled' in the study at the time of the BE Lead procedure.
Groups:
- Basic Evaluation Subjects: Out of 134 overactive bladder consented subjects in the study, 110 underwent basic evaluation with the commercially approved foramen needle and basic evaluation kit, and 107 subjects completed the study.
Period: Overall Study
Arm/Group | Basic Evaluation Subjects
Started | 110
Completed | 107
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Subjects with overactive bladder who went through InterStim basic evaluation with the commercially approved foramen needle and basic evaluation kit (110) and who had baseline information collected, were included.
Groups:
- Baseline: Subjects with overactive bladder who went through InterStim basic evaluation with the commercially approved foramen needle and basic evaluation kit
Arm/Group | Baseline
Number analyzed (Participants) | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (14.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity was only collected for subjects in the US - was not collected for EU or Canada.
  Participants
    number analyzed (Participants) | 75
    Hispanic or Latino | 7
    Not Hispanic or Latino | 68
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race was only collected for subjects in the US - was not collected for EU or Canada.
  Participants
    number analyzed (Participants) | 75
    American Indian or Alaska Native | 1
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 4
    White | 70
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Motor or Sensory Response(s) During Lead Placement - by Subject
Description: To characterize the proportion of subjects who demonstrate motor or sensory response(s) during lead placement using the InterStim basic evaluation lead.
  A motor or sensory response was determined at the time of lead placement. Amplitude was titrated up from 0 until a response was reported and/or observed. A sensory response was defined as the lowest amplitude where the subject first perceived sensation of the stimulation. A motor response was defined as the lowest amplitude of electrical stimulation where a motor response (e.g. bellows response, anal wink and/or plantar flexion of the big toe) was observed.
Time Frame: During lead implant procedure (approximately 20 minutes)
Population: Subjects with overactive bladder who went through InterStim basic evaluation with the commercially approved foramen needle and basic evaluation kit (110) were included.
Measure: Count of Participants; unit: Participants
Groups:
- Motor or Sensory Response of Lead: Response to Lead
- Motor or Sensory Response of Needle: Response to Needle
Arm/Group | Motor or Sensory Response of Lead | Motor or Sensory Response of Needle
Number analyzed (Participants) | 110 | 110
Participants
  Yes | 107 | 109
  No | 3 | 1

ADVERSE EVENTS:
Time Frame: From time of consent to one-week post lead placement
Description: All serious, device related, procedure-related, and/or therapy-related adverse events were considered reportable for this study
Groups:
- Basic Evaluation Subjects: For the mortality and serious adverse events, all consented subjects (134) were included. Since non-serious events can only be device, therapy or stimulation related, only subjects with overactive bladder who went through InterStim basic evaluation with the commercially approved foramen needle and basic evaluation kit (110) were included.
Arm/Group | Basic Evaluation Subjects
All-Cause Mortality (participants affected / at risk) | 0/134
Serious Adverse Events (participants affected / at risk) | 1/134
Other Adverse Events (participants affected / at risk) | 3/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Basic Evaluation Subjects (N=134)
Gastritis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Basic Evaluation Subjects (N=110)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT04016324/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT04016324/SAP_001.pdf